CLINICAL TRIAL: NCT00465023
Title: Phase I Study of Proton Beam Irradiation for the Treatment of Unresectable Hepatocellular Cancer or Hepatic Metastases
Brief Title: Proton Beam Irradiation for the Treatment of Unresectable Hepatocellular Cancer or Hepatic Metastases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Dana-Farber Cancer Institute (Other); Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Theodore Sunki Hong, Attending Radiation Oncologist, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-084
Record Dates: First submitted 2007-04-23; First posted 2007-04-24 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Hepatocellular Cancer; Cholangiocarcinoma; Hepatic Metastases
Keywords: proton beam irradiation; liver cancer
MeSH Terms: conditions — Liver Neoplasms; Cholangiocarcinoma | interventions — Proton Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Proton Beam Radiation (Experimental): Proton radiation therapy
  Interventions: Procedure: Proton Beam Radiation

INTERVENTIONS:
Procedure: Proton Beam Radiation — Once a day, 5 days a week (Monday-Friday) for 3 weeks.

SUMMARY:
The main purpose of this study is to determine if high doses of radiation using proton beam can be given safely with low and acceptable side effects. We will also gather information to determine the ability of proton beam to destroy cancer cells in the liver. There are two types of external radiation treatments (proton beam and photon beam). Proton beam radiation is a very accurate kind of treatment that has been shown to affect less normal tissue than a regular radiation beam. The accuracy allows us to more safely increase the amount of radiation delivered to eliminate cancer and may potentially reduce the side effects normally experienced with standard radiation therapy.

DETAILED DESCRIPTION:
* Participants will receive treatment as an outpatient at the Northeast Proton Treatment Center located at the Massachusetts General Hospital.
* Since we are looking for the highest dose of proton beam radiation that can be given to people safely, not everyone who participates in this study will be receiving the same amount of radiation. Small groups of people will be enrolled and given a certain dose of radiation. If they tolerate it well, the next small group of people enrolled will receive a higher dose. This will continue until we find the highest dose that can be given without causing serious or unmanageable side effects.
* Radiation treatment to the liver will be given once a day, 5 days a week (Monday-Friday), for 3 weeks. Each treatment takes about 10-20 minutes.
* A physical examination, medical history, and blood tests will be taken once a week for 3 weeks during radiation therapy. Follow-up visits will occur every 3 months for 2 years, and every 6 months thereafter for 3 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven unresectable or locally recurrent hepatocellular cancer, cholangiocarcinoma, or hepatic metastases.
* Primary lesion size of 6cm or less in greatest diameter
* Single or multinodular tumors (up to 3)
* 18 years of age or older
* No evidence of extrahepatic tumor
* Karnofsky performance status of 70-100
* If patient has underlying cirrhosis, only Child's classification Group A or Group B
* Adequate renal function
* Expected survival of greater than three months

Exclusion Criteria:

* Pregnant or lactating women
* Evidence of non-hepatic metastatic disease
* Local conditions or systemic illnesses which would reduce the local tolerance to radiation treatment, such as serious local injuries, active collagen vascular disease, etc.
* Prior radiation treatment to affected region
* Serious psychiatric illness which would limit compliance with treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2003-06; Primary Completion 2013-09 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) of proton beam irradiation in patients with unresectable or locally recurrent hepatocellular cancer, cholangiocarcinoma, or hepatic metastases. | 4 years

SECONDARY OUTCOMES:
To determine safety and tolerance of this treatment program | 4 years
to evaluate tumor response, local control and survival in this patient population.

CONTACTS AND LOCATIONS:
Overall Officials: Theodore S. Hong, MD, Principal Investigator — Massachusetts General Hospital